CLINICAL TRIAL: NCT00569127
Title: Phase III Prospective Randomized Comparison of Depot Octreotide Plus Interferon Alpha Versus Depot Octreotide Plus Bevacizumab (NSC #704865) in Advanced, Poor Prognosis Carcinoid Patients
Brief Title: Octreotide Acetate and Recombinant Interferon Alfa-2b or Bevacizumab in Treating Patients With Metastatic or Locally Advanced, High-Risk Neuroendocrine Tumor
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00778; NCI-2009-00778 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S0518; CDR0000579151; SWOG-S0518; S0518 (Other: SWOG); S0518 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Results first posted 2016-04-28 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Neuroendocrine Tumor G1; Gastric Neuroendocrine Tumor G1; Neuroendocrine Neoplasm; Neuroendocrine Tumor; Neuroendocrine Tumor G2
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Octreotide; Acetates; Salts; Introns; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (octreotide acetate and bevacizumab) (Experimental): Patients receive depot octreotide acetate IM and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Drug: Octreotide Acetate
- Arm II (octreotide acetate and recombinant interferon alfa-2b) (Experimental): Patients receive octreotide acetate IM as in arm I on day 1 and recombinant interferon alfa-2b SC on days 1, 3, 5, 8, 10, 12, 15, 17, and 19. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Octreotide Acetate; Biological: Recombinant Interferon Alfa-2b

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm I (octreotide acetate and bevacizumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Octreotide Acetate — Given IM
  Other Names: D-Phenylalanyl-L-cysteinyl-L-phenylalanyl-D-tryptophyl-L-lysyl-L-threonyl-N-[(1R,2R)-2-hydroxy-1-(hyroxymethyl)propyl]-L-cysteinamide, Cyclic (2->7)-disulfide, Acetate (Salt); Longastatin; Longastatina; Mycapssa; Samilstin; Sandostatin; Sandostatin LAR; Sandostatin Lar Depot; Sandostatina; Sandostatine; SMS 201-995; SMS 201-995 AC
Biological: Recombinant Interferon Alfa-2b — Given SC
  Other Names: Alfatronol; Bioferon; Bioferon (TM); Glucoferon; Heberon Alfa; IFN alpha-2B; Interferon alfa 2b; Interferon Alfa-2B; Interferon Alpha-2b; Intron A; Sch 30500; Urifron; Viraferon
  Arms: Arm II (octreotide acetate and recombinant interferon alfa-2b)

SUMMARY:
This randomized phase III trial studies octreotide acetate and recombinant interferon alfa-2b to see how well it works compared to octreotide acetate and bevacizumab in treating patients with high-risk neuroendocrine tumors that have spread to other places in the body (metastatic) or spread from where it started to nearby tissue or lymph nodes (locally advanced). Octreotide acetate and recombinant interferon alfa-2b may interfere with the growth of tumor cells and slow the growth of cancer. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. It is not yet known whether giving octreotide acetate together with recombinant interferon alfa-2b is more effective than giving octreotide acetate together with bevacizumab in treating patients with neuroendocrine tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare central review-based progression-free survival in poor prognosis carcinoid patients treated with either depot octreotide (octreotide acetate) plus bevacizumab, or depot octreotide plus interferon (recombinant interferon alfa-2b).

SECONDARY OBJECTIVES:

I. To compare overall survival, time to treatment failure and traditionally reported progression-free survival in poor prognosis carcinoid patients treated with either depot octreotide plus bevacizumab, or depot octreotide plus interferon.

II. To compare objective response (confirmed and unconfirmed complete response [CR] and partial response [PR]) in poor prognosis carcinoid patients treated with either depot octreotide plus bevacizumab, or depot octreotide plus interferon.

III. To compare the toxicity profile of patients treated with these two regimens.

TERTIARY OBJECTIVES:

I. To assess the prognostic and predictive value of vascular endothelial growth factor (VEGF) expression in relation to progression-free survival and treatment effect.

II. To compare response of 5HIAA, chromogranin A and neuronspecific enolase among patients with elevated levels at baseline between patients treated with octreotide plus interferon versus octreotide plus bevacizumab.

III. To assess and compare the prognostic and predictive value of the combination of In-111 pentetreotide somatostatin-receptor scintigraphy (SRS) and computed tomography (CT) vs. CT in relation to progression-free survival (PFS).

IV. To assess and compare the prognostic and predictive value of the combination of SRS and CT vs. CT in relation to overall survival (OS) and time to treatment failure (TTF).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive octreotide acetate intramuscularly (IM) and bevacizumab intravenously (IV) over 30-90 minutes on day 1.

ARM II: Patients receive octreotide acetate IM on day 1 and recombinant interferon alfa-2b subcutaneously (SC) on days 1, 3, 5, 8, 10, 12, 15, 17, and 19.

Treatment in both arms repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2-6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have unresectable metastatic or locally advanced, low- or intermediate-grade neuroendocrine carcinoma

  * NOTE: pathology report must state one of the following: carcinoid, low-grade or well-differentiated neuroendocrine carcinoma, atypical carcinoid, intermediate-grade or moderately differentiated neuroendocrine carcinoma; patients with poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid, or goblet cell carcinoid are not eligible; patient must not have osseous metastasis as only site of disease; patients with medullary thyroid carcinoma or islet cell carcinoma are not eligible; if pathology report states only neuroendocrine carcinoma, pathology subtype must be reconfirmed
  * Occasionally, it is not possible to establish tumor grade on fine-needle aspiration (FNA) cytology material; if a new biopsy is needed, a core needle biopsy should be obtained whenever possible
* Patient must have high risk disease as defined by at least one of the following:

  * Progressive disease
  * Refractory carcinoid syndrome while receiving octreotide (defined by > 2 flushing episodes/day or > 4 bowel movements/day)
  * Atypical histology and more than 6 lesions
  * Metastatic colorectal carcinoid; patients with metastatic cecal or appendiceal carcinoid tumor are not eligible unless the tumors fit into one of the other high-risk categories (a, b, or c above)
  * Metastatic gastric carcinoid
* Patient must have measurable disease; CT or magnetic resonance imaging (MRI) used for tumor measurement must have been completed within 28 days prior to registration; X-rays, scans or other tests for assessment of non-measurable disease must have been performed within 42 days prior to registration; all disease must be assessed and documented on the Baseline Tumor Assessment Form; these scans also must be submitted for central radiology review
* Institutions are required to submit CT/MRI scans and archived tissue for pathology review; furthermore, institutions are required to seek additional patient consent for submission of octreotide scans, and submission of blood and use of archived tissue for correlative studies
* If patient consents to the submission of octreotide scans, the patient must also be registered to Registration Step 2
* Patient may have had up to one prior regimen of cytotoxic chemotherapy; at least 28 days must have elapsed since completion of prior therapy, and patient must have recovered from all effects
* Patient may have had prior hepatic artery embolization; at least 28 days must have elapsed since embolization and there must be residual measurable disease; chemoembolization will be considered as one prior chemotherapy regimen
* Patient must not have received prior interferon, bevacizumab or any other therapy targeting VEGF or VEGF receptors
* Patient may have received prior therapy targeting stem cell factor receptor (c-kit), abelson murine leukemia viral oncogene homolog 1 (abl), platelet-derived growth factor receptor (PDGFR), mammalian target of rapamycin (mTOR), and somatostatin receptors (not counted toward prior cytotoxic chemotherapy)
* Prior radiation is allowed; there must be measurable disease; if prior therapies include peptide receptor radiotherapy, the target lesion(s) must have shown disease progression; at least 28 days must have elapsed since completion of prior therapy, and patient must have recovered from all effects
* Patients must have recovered from any prior surgery; one week must have elapsed from the time of a minor surgery and 4 weeks from major surgery
* At least 21 days must have elapsed since any prior octreotide LAR depot treatment
* Patient must have a Zubrod performance status of 0-2
* Absolute neutrophil count (ANC) > 1,500/mcl
* Hemoglobin > 8 g/dl
* Platelets > 100,000/mcl
* Serum bilirubin < 1.5 x institutional upper limit of normal (IULN)
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) =< 2.5 x IULN
* Serum creatinine < 1.5 mg/dL
* Urine protein must be screened by urine analysis for Urine Protein Creatinine (UPC) ratio; for UPC ratio > 0.5, 24-hour urine protein must be obtained and the level must be < 1,000 mg for patient enrollment; these results must be obtained within 28 days prior to registration

  * Note: UPC ratio of spot urine is an estimation of the 24-hour urine protein excretion - a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm
* Patients not on anticoagulation must have prothrombin time (PT) and partial thromboplastin time (PTT) =< 1.1 x lULN obtained within 28 days prior to registration; patients on full-dose anticoagulation (warfarin or low molecular weight heparin) are eligible provided that both of the following criteria are met:

  * The patient has an in-range international normalized ratio (INR) (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
  * The patient has no active bleeding or pathological condition that carries a high risk of bleeding such as varices
* Patient must not have history or evidence of clinically significant peripheral vascular disease such as non-healing peripheral ulcers or claudication
* Patient must not have a history of primary brain tumor or metastatic cancer to the brain; brain imaging studies are not required for eligibility if the patient has no neurological signs or symptoms; if brain imaging studies are performed, they must be negative for disease
* Patient must not have a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to registration
* Patient must not have history within the past 5 years or presence of bleeding diathesis or coagulopathy that results in spontaneous bleeding (in the absence of trauma) requiring packed red blood cells (pRBC) transfusion
* Patient must not have a serious (requiring active medical therapy with medication or medical device under the supervision of a physician) non-healing wound, ulcer, or bone fracture
* Patient must not have recent history (within 6 months prior to registration) of these arterial thromboembolic events: transient ischemic attack, cerebrovascular accident, unstable angina, myocardial infarction, or New York Heart Association grade II or higher congestive heart failure
* Patients with a history of hypertension must be well-controlled (blood pressure < 150/90), on a stable regimen of antihypertensive therapy
* Patient must not have hemoglobinopathies (e.g., Thalassemia) or any other cause of hemolytic anemia
* Patient must not plan to use any other concurrent chemotherapy, immunotherapy, hepatic artery embolization, hepatic artery chemoembolization, radiofrequency ablation, other tumor ablative procedure or radiotherapy while on protocol treatment
* Patient must not be pregnant or nursing because bevacizumab may be harmful to the developing fetus and newborn; male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout protocol treatment and for up to 6 months following discontinuation of bevacizumab
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, or any other cancer from which the patient has been disease free for five years
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and identification (ID) number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional re view board approval for this study has been entered into the data base
* REGISTRATION STEP 2 - SPECT SUBSTUDY
* Patient must have registered to the main study
* Patient must have consented to the submission of octreotide scans
* An octreotide scan obtained within 28 days prior to Registration Step 1 must be available for submission

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2007-12-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2026-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: James C Yao, Principal Investigator — SWOG Cancer Research Network
Locations (496):
- United States (496):
  - Providence Hospital, Mobile, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Arroyo Grande Community, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Sutter Cancer Research Consortium, Novato, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Montrose Memorial Hospital, Montrose, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - MacNeal Hospital and Cancer Center, Berwyn, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Saint Anthony Memorial Hospital, Effingham, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - MercyOne Genesis Davenport Cancer Center, Davenport, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Our Lady Bellefonte Hospital, Ashland, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center, Jackson, Mississippi
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Garnet Health Medical Center, Middletown, New York
  - Highland Hospital, Rochester, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Geisinger South Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - NCORP of the Carolinas (Prisma Health NCORP), Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Tennessee Cancer Specialists-Dowell Springs, Knoxville, Tennessee
  - East Tennessee Baptist Hospital-Mercy Health Partners, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Yao JC, Guthrie KA, Moran C, Strosberg JR, Kulke MH, Chan JA, LoConte N, McWilliams RR, Wolin EM, Mattar B, McDonough S, Chen H, Blanke CD, Hochster HS. Phase III Prospective Randomized Comparison Trial of Depot Octreotide Plus Interferon Alfa-2b Versus Depot Octreotide Plus Bevacizumab in Patients With Advanced Carcinoid Tumors: SWOG S0518. J Clin Oncol. 2017 May 20;35(15):1695-1703. doi: 10.1200/JCO.2016.70.4072. Epub 2017 Apr 6. PMID 28384065
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Octreotide, Bevacizumab: Patients receive 20 mg depot octreotide acetate IM and 15 mg/kg bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
- Octreotide, Interferon Alpha-2b: Patients receive 20 mg depot octreotide acetate IM on day 1 and 5 million units interferon alpha-2b three times per week (Days 1, 3, 5, 8, 10, 12, 15, 17, 19 of each cycle). Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Octreotide, Bevacizumab | Octreotide, Interferon Alpha-2b
Started | 214 | 213
Eligible | 200 | 202
Completed | 0 | 0
Not Completed | 214 | 213
Not completed — Adverse Event | 57 | 47
Not completed — Withdrawal by Subject | 13 | 27
Not completed — Progression | 99 | 100
Not completed — Death | 4 | 3
Not completed — Other | 20 | 19
Not completed — Lost to Follow-up | 0 | 3
Not completed — Not Eligible | 14 | 11
Not completed — Still on Treatment | 7 | 3

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Octreotide, Bevacizumab | Octreotide, Interferon Alpha-2b | Total
Number analyzed (Participants) | 200 | 202 | 402
Age, Continuous [Median (Full Range); unit: years] | 60.5 [27.2 to 85.3] | 61.1 [23.1 to 85.4] | 60.9 [23.1 to 85.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 112 | 210
  Male | 102 | 90 | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 11 | 24
  Not Hispanic or Latino | 166 | 177 | 343
  Unknown or Not Reported | 21 | 14 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 18 | 20 | 38
  White | 169 | 167 | 336
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 3 | 11 | 14
Disease Site [Number; unit: participants]
  Small bowel, cecum, appendix | 71 | 72 | 143
  Other sites | 129 | 130 | 259
Progression after Initial Diagnosis [Number; unit: participants]
  Yes | 182 | 188 | 370
  No | 18 | 14 | 32
Histologic Grade [Number; unit: participants]
  Low | 169 | 171 | 340
  Intermediate (atypical) | 31 | 31 | 62
Prior Octreotide [Number; unit: participants]
  Within 2 months prior to registration | 114 | 115 | 229
  None within 2 months prior to registration | 86 | 87 | 173

OUTCOME MEASURES:

1. Secondary Outcome: Overall Survival
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Up to 7 years
Population: According to the intent-to-treat principle, all eligible patients will be included in this analysis according to the randomized treatment assignment, regardless of actual treatments received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Octreotide, Bevacizumab | Octreotide, Interferon Alpha-2b
Number analyzed (Participants) | 200 | 202
months | 35.2 [33.1 to 42.8] | 47.3 [35.8 to 52.6]

2. Primary Outcome: Central Review-based Progression-Free Survival
Description: From date of randomization (which is the date of registration) to date of first documentation of progression based on Central Radiological Review of the appropriate CT or MRI scans, or symptomatic deterioration (as defined in Section 10.2e)), or development of new lesions or disease not identified on CT or MRI, or death due to any cause. Patients who have a local assessment of progression based on imaging, but for whom central review does not concur, will be censored at the last Central Radiological Review date, unless subsequent scans or documentation of symptomatic deterioration provides evidence of progression. Patients last known not to have progressed are censored at the date of last contact. Patients with incomplete Central Radiological Review are censored at the date of last Central Radiological Review if patient has not progressed prior to that time.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Octreotide, Bevacizumab | Octreotide, Interferon Alpha-2b
Number analyzed (Participants) | 200 | 202
months | 16.6 [12.9 to 19.6] | 15.4 [9.6 to 18.6]
Statistical Analysis 1: Comparison: Octreotide, Bevacizumab vs Octreotide, Interferon Alpha-2b; According to the intent-to-treat principle, all eligible patients were included in the analysis according to the randomized treatment assignment, regardless of actual treatments received; Test type: Superiority or Other; p = 0.55, Regression, Cox — Central-review based progression-free survival was analyzed using the stratified log rank test (which is the score test from the stratified Cox-model) using stratification factors as defined in Section 6.0; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.73 to 1.18] — The reported hazard ratio estimate is for the comparison of the Octreotide, Bevacizumab arm to the Octreotide, Interferon Alpha-2b arm

3. Secondary Outcome: Time to Treatment Failure
Description: From date of randomization (which is the date of registration) to date of first observation of progressive disease (as defined in Section 10.2d), death due to any cause, symptomatic deterioration (as defined in Section 10.2e), or discontinuation of treatment. This has been calculated using Central-Review based progression events. Patients last known not to have failed treatment are censored at date last known not to have failed. Patients with incomplete Central Radiological Review are censored at the date of last Central Radiological Review if patient has not failed treatment prior to that time.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Octreotide, Bevacizumab | Octreotide, Interferon Alpha-2b
Number analyzed (Participants) | 200 | 202
months | 9.9 [7.3 to 11.1] | 5.6 [4.3 to 6.4]

4. Secondary Outcome: Local Progression-Free Survival (Investigator Assessed)
Description: From date of randomization (which is the date of registration) to date of first documentation of progression [per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) as defined in Section 10.2d] or symptomatic deterioration (as defined in Section 10.2e), or death due to any cause. Patients last known not to have progressed are censored at date of last contact. Progression (Section 10.2d) includes one or more of the following: 20% increase in the sum of the longest diameters of target measurable lesions over smallest sum observed using the same techniques as baseline; unequivocal progression of non-measurable disease in the opinion of the treating physician; appearance of new lesion/site; or death due to disease without prior documentation of progression and without symptomatic deterioration. Symptomatic deterioration (Section 10.2e) is global deterioration of health status requiring discontinuation of treatment without objective evidence of progression.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Octreotide, Bevacizumab | Octreotide, Interferon Alpha-2b
Number analyzed (Participants) | 200 | 202
months | 15.4 [12.6 to 17.2] | 10.6 [8.5 to 14.4]

5. Secondary Outcome: Objective Response (Confirmed and Unconfirmed Complete Response and Partial Response)
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0): Complete Response (CR) is disappearance of all measurable and non-measurable disease, and no new lesions; Partial Response (PR) is greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions, no unequivocal progression of non-measurable disease, and no new lesions. Confirmed response is two or more objective statuses of CR a minimum of four weeks apart documented before progression or symptomatic deterioration. Partial response is two or more objective statuses of PR or better a minimum of four weeks apart documented before progression or symptomatic deterioration. Unconfirmed CR is one objective status of CR documented before progression or symptomatic deterioration but not qualifying as CR or PR. Unconfirmed PR is one objective status of PR documented before progression or symptomatic deterioration but not qualifying as CR, PR or unconfirmed CR.
Time Frame: Up to 3 years
Population: All eligible patients with measurable disease will be included in this analysis according to the randomized treatment assignment.
Measure: Number; unit: participants
Arm/Group | Octreotide, Bevacizumab | Octreotide, Interferon Alpha-2b
Number analyzed (Participants) | 200 | 202
participants
  Complete Response | 2 | 0
  Partial Response | 20 | 8
  Unconfirmed Complete Response | 0 | 1
  Unconfirmed Partial Response | 7 | 6
  Stable/No Resposne | 135 | 137
  Increasing Disease | 20 | 30
  Symptomatic Deterioration | 0 | 3
  Assessment Inadequate | 16 | 17

6. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 3 years
Population: Eligible patients who received any treatment and were assessed for adverse events are included in this summary. Eleven patients did not start protocol treatment due to: patient refusal (6), financial reasons (3), and worsening condition/progression (2). None were assessable for adverse events and thus are not included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Octreotide, Bevacizumab | Octreotide, Interferon Alpha-2b
Number analyzed (Participants) | 197 | 194
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 0 | 4
  AST, SGOT | 1 | 6
  Albumin, serum-low (hypoalbuminemia) | 0 | 1
  Alkaline phosphatase | 2 | 6
  Allergic reaction/hypersensitivity | 1 | 0
  Anorexia | 1 | 8
  Ataxia (incoordination) | 2 | 0
  Auditory/Ear-Other (Specify) | 0 | 1
  Bilirubin (hyperbilirubinemia) | 1 | 1
  CNS cerebrovascular ischemia | 1 | 0
  Cardiac troponin I (cTnI) | 1 | 0
  Cardiac-ischemia/infarction | 1 | 0
  Cardiopulmonary arrest, cause unknown (non-fatal) | 0 | 1
  Cholecystitis | 2 | 0
  Cognitive disturbance | 1 | 1
  Colitis | 1 | 0
  Constipation | 1 | 1
  Creatinine | 1 | 0
  Dehydration | 3 | 5
  Dental: periodontal disease | 1 | 0
  Diarrhea | 7 | 9
  Dizziness | 2 | 3
  Dyspnea (shortness of breath) | 1 | 2
  Edema: limb | 4 | 1
  Fatigue (asthenia, lethargy, malaise) | 13 | 50
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 0 | 1
  Fistula, GI - Colon/cecum/appendix | 1 | 0
  Fistula, GU - Vagina | 1 | 0
  Glucose, serum-high (hyperglycemia) | 2 | 5
  Hearing: pts w/o audiogram not enroll monitor prgm | 0 | 1
  Heartburn/dyspepsia | 1 | 0
  Hemoglobin | 0 | 4
  Hemorrhage, CNS | 2 | 0
  Hemorrhage, GI - Rectum | 1 | 0
  Hemorrhage, GI - Upper GI NOS | 1 | 0
  Hemorrhage, pulmonary/upper respiratory - Nose | 1 | 0
  Hemorrhage/Bleeding-Other (Specify) | 1 | 0
  Hot flashes/flushes | 0 | 1
  Hydrocephalus | 1 | 0
  Hypertension | 62 | 4
  Hypotension | 2 | 0
  Hypoxia | 1 | 0
  INR (of prothrombin time) | 1 | 0
  Ileus, GI (functional obstruction of bowel) | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Nose | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Ab NOS | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 2 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 1 | 2
  Infection with unknown ANC - Scrotum | 1 | 0
  Infection with unknown ANC - Urinary tract NOS | 1 | 0
  Insomnia | 0 | 1
  Left ventricular systolic dysfunction | 1 | 0
  Leukocytes (total WBC) | 2 | 14
  Lipase | 0 | 1
  Lymphopenia | 3 | 5
  Mental status | 1 | 1
  Mood alteration - agitation | 0 | 2
  Mood alteration - anxiety | 0 | 1
  Mood alteration - depression | 1 | 7
  Mucositis/stomatitis (clinical exam) - Oral cavity | 0 | 1
  Mucositis/stomatitis (functional/symp) - Oral cav | 1 | 0
  Muscle weakness, not d/t neuropathy - body/general | 0 | 3
  Nausea | 5 | 9
  Neuropathy: motor | 1 | 1
  Neutrophils/granulocytes (ANC/AGC) | 0 | 23
  Obstruction, GI - Gallbladder | 1 | 0
  Obstruction, GI - Small bowel NOS | 2 | 1
  Pain - Abdomen NOS | 7 | 5
  Pain - Back | 1 | 2
  Pain - Bone | 0 | 1
  Pain - Chest wall | 2 | 1
  Pain - Chest/thorax NOS | 2 | 2
  Pain - Esophagus | 1 | 0
  Pain - Extremity-limb | 1 | 1
  Pain - Gallbladder | 0 | 1
  Pain - Head/headache | 9 | 3
  Pain - Liver | 0 | 1
  Pain - Muscle | 1 | 1
  Pain - Stomach | 0 | 1
  Pain-Other (Specify) | 1 | 1
  Phosphate, serum-low (hypophosphatemia) | 1 | 0
  Platelets | 3 | 0
  Pneumonitis/pulmonary infiltrates | 1 | 1
  Potassium, serum-low (hypokalemia) | 1 | 1
  Proteinuria | 17 | 1
  Pruritus/itching | 0 | 1
  Rash/desquamation | 1 | 1
  Renal failure | 0 | 1
  Renal/Genitourinary-Other (Specify) | 2 | 0
  Seizure | 0 | 2
  Sodium, serum-low (hyponatremia) | 1 | 0
  Somnolence/depressed level of consciousness | 3 | 1
  Syncope (fainting) | 2 | 1
  Thrombosis/embolism (vascular access-related) | 3 | 1
  Thrombosis/thrombus/embolism | 3 | 1
  Triglyceride, serum-high (hypertriglyceridemia) | 0 | 1
  Ulcer, GI - Duodenum | 1 | 0
  Ulcer, GI - Stomach | 1 | 0
  Uric acid, serum-high (hyperuricemia) | 1 | 0
  Vasculitis | 0 | 1
  Vessel injury-artery - Aorta | 1 | 0
  Vision-blurred vision | 0 | 1
  Vomiting | 4 | 2
  Weight loss | 2 | 3

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Eligible patients who received treatment and were assessed for adverse events are included in the adverse event summaries. Eleven patients did not start protocol treatment due to: patient refusal (6), financial reasons (3), and worsening condition/progression (2). None were assessable for adverse events and thus are not included in this analysis.
Arm/Group | Octreotide, Bevacizumab | Octreotide, Interferon Alpha-2b
Serious Adverse Events (participants affected / at risk) | 68/197 | 9/194
Other Adverse Events (participants affected / at risk) | 103/197 | 98/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide, Bevacizumab (N=197) | Octreotide, Interferon Alpha-2b (N=194)
Hemoglobin (Blood and lymphatic system disorders) | 2 | 0
Cardiac Arrhythmia-Other (Cardiac disorders) | 1 | 0
Cardiac General-Other (Cardiac disorders) | 1 | 0
Cardiac-ischemia/infarction (Cardiac disorders) | 1 | 0
Cardiopulmonary arrest, cause unknown (non-fatal) (Cardiac disorders) | 0 | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 | 0
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1 | 0
Ascites (non-malignant) (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Distention/bloating, abdominal (Gastrointestinal disorders) | 1 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2 | 0
Esophagitis (Gastrointestinal disorders) | 2 | 0
Fistula, GI - Colon/cecum/appendix (Gastrointestinal disorders) | 1 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 1 | 0
Ileus, GI (functional obstruction of bowel) (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 7 | 0
Obstruction, GI - Colon (Gastrointestinal disorders) | 2 | 0
Obstruction, GI - Ileum (Gastrointestinal disorders) | 1 | 0
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 8 | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 17 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Perforation, GI - Colon (Gastrointestinal disorders) | 1 | 0
Perforation, GI - Small bowel NOS (Gastrointestinal disorders) | 1 | 1
Ulcer, GI - Duodenum (Gastrointestinal disorders) | 1 | 0
Ulcer, GI - Jejunum (Gastrointestinal disorders) | 1 | 0
Ulcer, GI - Stomach (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Death not associated with CTCAE term - Death NOS (General disorders) | 1 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 | 1
Pain - Chest/thorax NOS (General disorders) | 2 | 0
Pain-Other (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Obstruction, GI - Gallbladder (Hepatobiliary disorders) | 1 | 0
Allergic reaction/hypersensitivity (Immune system disorders) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Ab NOS (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Bladder (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 1 | 0
Infection with unknown ANC - Blood (Infections and infestations) | 2 | 0
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 2 | 0
Infection with unknown ANC - Scrotum (Infections and infestations) | 1 | 0
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1 | 0
Infection with unknown ANC - Wound (Infections and infestations) | 1 | 0
Vessel injury-artery - Aorta (Injury, poisoning and procedural complications) | 1 | 0
AST, SGOT (Investigations) | 1 | 0
Alkaline phosphatase (Investigations) | 1 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 1 | 1
CD4 count (Investigations) | 1 | 0
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 0 | 1
Cardiac troponin I (cTnI) (Investigations) | 1 | 0
Creatinine (Investigations) | 1 | 0
Lymphopenia (Investigations) | 2 | 0
Platelets (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 9 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 | 0
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 | 0
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 | 1
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Secondary Malignancy-poss rel to cancer Tx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (incoordination) (Nervous system disorders) | 1 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Hemorrhage, CNS (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Pain - Head/headache (Nervous system disorders) | 5 | 0
Somnolence/depressed level of consciousness (Nervous system disorders) | 3 | 0
Syncope (fainting) (Nervous system disorders) | 3 | 0
Confusion (Psychiatric disorders) | 2 | 0
Mood alteration - depression (Psychiatric disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 4 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal/Genitourinary-Other (Renal and urinary disorders) | 1 | 0
Fistula, GU - Vagina (Reproductive system and breast disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 5 | 0
Hypotension (Vascular disorders) | 4 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide, Bevacizumab (N=197) | Octreotide, Interferon Alpha-2b (N=194)
Diarrhea (Gastrointestinal disorders) | 16 | 13
Nausea (Gastrointestinal disorders) | 8 | 13
Pain - Abdomen NOS (Gastrointestinal disorders) | 17 | 17
Fatigue (asthenia, lethargy, malaise) (General disorders) | 19 | 55
Leukocytes (total WBC) (Investigations) | 5 | 14
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2 | 23
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 8 | 14
Pain - Back (Musculoskeletal and connective tissue disorders) | 5 | 10
Proteinuria (Renal and urinary disorders) | 14 | 1
Hypertension (Vascular disorders) | 60 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less